CLINICAL TRIAL: NCT01060618
Title: Estudio Comparativo de Dos métodos Para Predecir el Uso de Co-receptores Por el Virus de la Inmunodeficiencia 1 (HIV-1): el Ensayo fenotípico (Trofile ESTA®) y la Respuesta virológica a Corto Plazo a un Antagonista de CCR5
Brief Title: Double-method Comparative Study in Order to Predict the Use of Co-receptors From Type 1 HIV: Phenotypic Study (Trofile ESTA®) and Virologic Response to a CCR5 Antagonist in the Short Term
Acronym: TROPISMVC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TROPISMVC; 2008-007208-28 (Other: EudraCT Number (EMEA))
Record Dates: First submitted 2010-01-31; First posted 2010-02-02 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maraviroc + Trofile ESTA® (Experimental): the patients have the Trofile ESTA® test performed and sent for evaluation. Once the results are obtained (about 1 month later), the patients take the medication Maraviroc during ten days. The viral load assessment throughout the Study help to make a prediction to assess if the patients would have a positive response Vs. CCR5 antagonist of a negative response
  Interventions: Other: Maraviroc + Trofile ESTA® (diagnose test)

INTERVENTIONS:
Other: Maraviroc + Trofile ESTA® (diagnose test) — The Trofile ESTA® will be performed in those patients and once the results are obtained (within one month approximately), the patients will be treated with the medication Maraviroc

SUMMARY:
The summary of the Study is to compare two methods in order to predict how the 1-HIV will use a co-receptor: the use of an accredited test (TROFILE ESTA®) and the viral response to a CCR5 antagonist in the short term.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to give, sign and date the Informed Consent Form to participate in the Study and to donate their samples for cell and molecular Studies, after receiving the appropriate information about the Study design, the main objective of the Study and the potential risks.
* Patients aged >18.
* Patients with chronic HIV infection
* Patients with no previous HAART (naïve patients).
* Patients that do not meet HAART starting criteria.
* Viral load >1.000 HIV RNA copies/mL
* Patients able to understand the Study objectives and able to perform frequent visits to the Study Site.

Exclusion Criteria:

* Prior HAART (regardless of the HAART type).
* Pregnancy or willingness to get pregnant during the Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine if there is a correlation between the Trofile ESTA® test for viral tropism and the viral load reduction after a short treatment with maraviroc in naïve patients (patients with no previous HAART) | 10 days of treatment per patient

SECONDARY OUTCOMES:
To establish a viral load reduction cut point, which would differentiate R5-tropic virus from non-R5 tropic virus(X4/dual/mixed). | 1 month per patient
To assess the viral response to a CCR5 antagonist according to the viral tropism identified in the phenotypic Study. | 1 month per patient
Safety assessment throughout the Study | 12 months
Maraviroc effects assessment in the drug-resistance evolution in naïve patients | 12 months
Tropism changes assessment since the Screening period | 1 month per patient

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Moreno, MD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (4):
- Spain (4):
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid

REFERENCES:
- [Derived] Cascajero A, Rastrojo A, Diez-Fuertes F, Hernandez-Novoa B, Aguado B, Moreno S, Alcami J, Perez-Olmeda M. Deep-Sequencing Analysis of the Dynamics of HIV-1 Quasiespecies in Naive Patients during a Short Exposure to Maraviroc. J Virol. 2018 May 14;92(11):e00390-18. doi: 10.1128/JVI.00390-18. Print 2018 Jun 1. PMID 29563289
- [Derived] Hernandez-Novoa B, Madrid-Elena N, Dronda F, Perez-Elias MJ, Casado JL, Perez-Molina JA, Moreno A, Estebanez M, Gonzalez J, Zamora J, Moreno S. Virological response to short-course maraviroc monotherapy does not predict viral tropism in HIV-1-infected treatment-naive patients. J Antimicrob Chemother. 2014 Jul;69(7):1916-9. doi: 10.1093/jac/dku059. Epub 2014 Mar 12. PMID 24623833